CLINICAL TRIAL: NCT01800682
Title: A Single-Dose, Open-Label, Randomized, Crossover Dose-Proportionality Study to Evaluate the Effect of Dose on the Pharmacokinetics of 25, 50, and 100 mg ULTRAM ER Under Fasted Conditions in Healthy Adult Subjects
Brief Title: A Pharmacokinetic Study to Evaluate the Dose-Proportionality of Tramadol (ULTRAM) Extended-Release (ER) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR018658; TRAM-PAI-1001
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Healthy; Tramodol; Ultram
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tramodol Extended-release (ER), 25 milligram (mg) (Experimental): Tramodol ER, 25 mg tablets will be administered orally once daily on Day 1 of each treatment period (separated with washout period of 4-14 days).
  Interventions: Drug: Tramodol Extended-Release (ER)
- Tramodol ER, 50 mg (Experimental): Tramodol ER, 50 mg tablets will be administered orally once daily on Day 1 of each treatment period (separated with washout period of 4-14 days).
  Interventions: Drug: Tramodol Extended-Release (ER)
- Tramodol ER, 100 mg (Experimental): Tramodol ER, 100 mg tablets will be administered orally once daily on Day 1 of each treatment period (separated with washout period of 4-14 days).
  Interventions: Drug: Tramodol Extended-Release (ER)

INTERVENTIONS:
Drug: Tramodol Extended-Release (ER) — Tramodol ER, will be administered orally as either 25, 50 or 100 milligram tablet, once daily on Day 1 of each treatment period (separated with washout period of 4-14 days).
  Other Names: - Ultram

SUMMARY:
The purpose of this study is to evaluate the dose proportionality of the pharmacokinetics (explores what the body does to the drug) of tramadol in healthy adult participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center, randomized (study drug assigned by chance), and 3-way crossover (method used to switch participants from one study group to another in a clinical trial) study of tramadol extended-release (ER). All participants will be randomly assigned to 1 of 6 possible treatment sequences of tramadol. The study consists of 3 parts: Screening (within 20 days before study commences on Day -1); Open-label treatment (consisting of 3 single-dose treatment periods separated with washout period of 4-14 days, and dosing will be under fasting conditions on Day 1 in each treatment period); and Follow-up (up to 48-hour blood sample collection on Day 3 of Period 3). The duration of study is anticipated to be 6-8 weeks per participant. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Females with negative pregnancy test at Screening and on Day -1 of each treatment period
* Postmenopausal Females (no spontaneous menses for at least 2 years), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control
* Body mass index (BMI; weight in kilogram [kg] divided by height in square meter [m^2]) from 18 to 30 kilogram per square meter (kg/m^2), and body weight not less than 50 kg
* Blood pressure (after the participant is supine for 5 minutes - average of a minimum of 2 readings taken at intervals of at least 1 minute) between 90 and 140 millimeter of mercury (mmHg) systolic (top number in blood pressure, pressure during active contraction of the heart), and no higher than 90 mmHg diastolic (lower number in blood pressure reading pertaining to resting or relaxation phase of heart beat)
* Non-Smoker

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospasmic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for laboratory tests at Screening
* Clinically significant abnormal physical examination, vital signs or electrocardiogram at Screening
* Use of any prescription or non-prescription medication (including monoamine oxidase inhibitors, laxatives, vitamins, and herbal supplements), except for acetaminophen, oral contraceptives and hormonal replacement therapy within 30 days before the first dose of the study drug is scheduled
* History of drug or alcohol abuse within the past 5 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of Tramadol | Predose and at 0, 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 15, 16, 20, 24, 36, and 48 hours post dose of study treatment
  The Cmax is the maximum plasma concentration.
Time to reach maximum concentration (tmax) of Tramadol | Predose and at 0, 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 15, 16, 20, 24, 36, and 48 hours post dose of study treatment
  The Tmax is time to reach the maximum plasma concentration.
Area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration (AUC[last]) | Predose and at 0, 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 15, 16, 20, 24, 36, and 48 hours post dose of study treatment
  The AUC(last) is the area under the plasma concentration-time curve from time 0 to time of the last quantifiable concentration.
Area under the plasma concentration-time curve from time 0 to infinite time (AUC[infinity]) | Predose and at 0, 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 15, 16, 20, 24, 36, and 48 hours post dose of study treatment
  The AUC(infinity) is the area under the plasma concentration-time curve from time 0 to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Elimination half-life period (t1/2) associated with the terminal slope (Lambda z) | Predose and at 0, 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 15, 16, 20, 24, 36, and 48 hours post dose of study treatment
  Elimination half-life associated with the terminal slope (lambda[z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Terminal slope (Lambda z) | Predose and at 0, 1, 2, 3, 4, 6, 8, 10, 12, 13, 14, 15, 16, 20, 24, 36, and 48 hours post dose of study treatment
  Terminal slope is defined by first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Overland Park, Kansas, United States